CLINICAL TRIAL: NCT04803942
Title: Clinical Intuition for PRedicting Evolution in Sepsis in the Emergency Department - CIPRES-ED Study
Acronym: CIPRES-ED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2020/S2/06
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Sepsis
Keywords: Sepsis; clinical intuition; emergency department
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sepsis is a syndrome involving infection and an abnormal systemic inflammatory response in the infected organism, resulting in organ dysfunction and possibly death. It is a major cause of hospital mortality. A large proportion of sepsis diagnoses are made in emergency departments. Early diagnosis and appropriate treatment have been shown to reduce mortality from this disease.

In a context of limited resources, it is therefore important to be able to quickly stratify patients presenting to the emergency department with a suspected infection into those who require rapid and intensive management because they are at risk of developing sepsis and septic shock and those who can be managed conventionally The objective of this study is to compare the clinical intuition of emergency room physicians and nurses with the qSOFA score to predict the clinical course of patients presenting to the emergency room with potential sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to one of the participating emergency departments with suspected infection, defined as the presence of at least one of these parameters:

Temperature ≥ 38°C ou < 36°C measured in the emergency room Chills (in the emergency room or on recent history)

* No objection to participation in the study

Exclusion Criteria:

* Minor patient (<18 years)
* Patient under guardianship or other protective measure
* Patient unable to understand research information
* Patient refusing the use of their data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to one of the participating emergency departments with suspected infection
Sampling Method: Non-Probability Sample
Enrollment: 692 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Compare emergency physicians' clinical intuition versus qSOFA score for prediction of 30-day mortality in patients with suspected infection | 1 month after inclusion
  We compare the area under the ROC curve of each test (Emergency physicians' clinical intuition versus qSOFA score) to predict 30-day mortality in patients with suspected infection

SECONDARY OUTCOMES:
Compare emergency physicians' clinical intuition versus qSOFA score for prediction of 72 hours mortality in patients with suspected infection | 72 hours after inclusion
  We compare the area under the ROC curve of each test (Emergency physicians' clinical intuition versus qSOFA score) to predict 72 hours mortality in patients with suspected infection

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France